CLINICAL TRIAL: NCT04960059
Title: NOTION: iN-home Sampling Of cyTokines in ImmunOtherapy patieNts
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp181
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Cancer; Metastatic Melanoma; Renal Cell Carcinoma; Non-small Cell Lung Cancer
Keywords: Immunotherapy; immune related adverse event; cytokine release
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
This study will explore the ability of patients on first line combination immunotherapy to sample cytokines at home. The data from this study will be used to evaluate the feasibility of in-home testing and the ability to analyse patients cytokine profiles retrospectively to help feed the development of further studies.

DETAILED DESCRIPTION:
Patients will be informed of the study and given a minimum of 24 hours to consider. Once consented patients will enter the study where they will take cytokine samples at home over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent.
* Aged at least 18 years.
* Diagnosis of locally advanced or metastatic RCC, Melanoma or NSCLC
* In the opinion of the investigator deemed suitable to receive first-line combination immunotherapy (RCC and MM) or combination immunotherapy and chemotherapy (NSCLC).
* Willingness to comply with scheduled trial procedures.
* Capable of performing own dry blood sampling procedure, or a carer who is willing and able to perform them.

Exclusion Criteria:

* Previous immunotherapy (including any CPI either as single agent on in combination, or high dose interleukin-2).
* Judgement by the investigator that the individual should not participate if they are unlikely to comply with study procedures and requirements.
* Patients receiving long term oral anticoagulation deemed by the clinician to be at risk from daily finger pricking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving checkpoint inhibitor therapy as first line treatment of renal cell carcinoma, metastatic melanoma or non-small cell lung cancer (in combination with chemotherapy for NSCLC).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient adherence to protocol defined DBS time points. | 12 months
  the number of DBS samples successfully collected against the number of total expected samples
Number of in-home DBS samples passing quality assurance checks in patients receiving CPI therapy by multi-cytokine ELISA. | 12 months
  the number of DBS samples passing quality assurance checks against the number of DBS samples successfully collected.

SECONDARY OUTCOMES:
Compare cytokine concentrations by DBS sampling and intravenous blood sampling by multi-cytokine ELISA. | 12 months
  The changes of cytokine concentrations will be estimated by the log-ratio of cytokine concentrations measured at two time points. The trend of cytokine concentration during treatment will be estimated by fitting a linear regression model based on all cytokine concentrations collected during treatment.

OTHER OUTCOMES:
Retrospective mapping of immune-related adverse events with cytokine concentrations over time by in-home DBS sampling. | 12 months
  The association between these statistics and the development of immune-related adverse events will be estimated using a logistic regression analysis.
Patient reported outcomes from semi-structured interviews. | 12 months
  The patient satisfaction level will be assessed by survey interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Graham, MD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No